CLINICAL TRIAL: NCT01118156
Title: Suicide Classification System
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Lisa A. Brenner, Ph.D., ABBP, Denver VA Medical Center
Other Study IDs: 09-0641
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Suicide and Self-harm
Keywords: Suicide Nomenclature
MeSH Terms: conditions — Suicide; Self-Injurious Behavior | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mental Health Clinicians: MH Clinicians at the Denver and Grand Junction VA Medical Centers
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — 75-minute training teaching utilization of new standardized suicide nomenclature
  Other Names: Nomenclature Training

SUMMARY:
The purpose of this study is to evaluate whether a new standardized language for categorizing suicidal and self-injury related thoughts and behaviors can be readily adopted for use by mental health clinicians. Efforts also include developing a measure that can be used to help clinicians identify appropriate terms (e.g., behaviors) for specific patients.

DETAILED DESCRIPTION:
In recent years, suicide prevention has received increased focus within the VA. This is in part related to concerns regarding the mental health and associated suicide risk of Operation Enduring Freedom/Operation Iraqi Freedom military personnel, and a recent study highlighting the increased risk of death by suicide for members of the veteran population. Suicide prevention initiatives could be greatly enhanced if a clinically feasible uniform language regarding suicidality and self-injury was readily available and adopted throughout the VA system. With this goal in mind, the Self-Directed Violence Classification System (SDVCS) and Clinical Tool were developed based upon the Centers for Disease Control and Prevention (CDC) nomenclature and VA VISN-19 MIRECC's work in this area. The purpose of this study is to evaluate whether a new standardized language for categorizing suicidal and self-injury related thoughts and behaviors can be readily adopted for use by mental health clinicians. Efforts also include developing a measure that can be used to help clinicians identify appropriate terms (e.g., behaviors) for specific patients.

ELIGIBILITY:
Inclusion Criteria:

* Suicide Prevention Coordinator team members at Denver or Grand Junction VA Medical Center
* Mental Health leadership at Denver or Grand Junction VA Medical Center
* Mental Health professionals at Denver or Grand Junction VA Medical Center

Exclusion Criteria:

* Failure to sign appropriate informed consent
* MIRECC staff members

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mental Health professionals at the Denver and Grand Junction VA Medical Centers
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Proportion of clinicians utilizing nomenclature | 6 months
  Clinician chart notes will be reviewed to determine use of standardized nomenclature. Among those clinicians utilizing the nomenclature, accurate use will also be assessed.

SECONDARY OUTCOMES:
Analysis of qualitative focus group data | 6 months
  Qualitative evaluation of organizational- and provider-level factors associated with implementation

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, PhD, Principal Investigator — VA ECHCS VISN 19 MIRECC
Locations (2):
- United States (2):
  - Denver VA Medical Center, Denver, Colorado
  - Grand Junction VA Medical Center, Grand Junction, Colorado

REFERENCES:
- See also: brief descriptions of current research at the VISN 19 MIRECC — http://www.mirecc.va.gov/visn19/